CLINICAL TRIAL: NCT04195893
Title: Refitting Frequent Replacement Lens Wearers Into Clariti 1 Day And 1-Day Acuvue Moist Daily Disposable Spherical Lenses (BEAGLE 2)
Brief Title: Refitting Frequent Replacement Lens Wearers Into Clariti 1 Day And 1-Day Acuvue Moist Daily Disposable Spherical Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-112
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- somofilcon A (Experimental): Subjects will be randomized to wear somofilcon A daily disposable lenses for one week and then switch to etafilcon A daily disposable lenses for one week.
  Interventions: Device: somofilcon A
- etafilcon A (Active Comparator): Subjects will be randomized to wear etafilcon A daily disposable lenses for one week and then switch to somofilcon A daily disposable lenses for one week.
  Interventions: Device: etafilcon A

INTERVENTIONS:
Device: somofilcon A — Contact Lens
  Other Names: Clariti 1-Day
  Arms: somofilcon A
Device: etafilcon A — Contact Lens
  Other Names: 1-Day Acuvue Moist
  Arms: etafilcon A

SUMMARY:
The objective of the study is to evaluate and compare the performance of somofilcon A to etafilcon A when worn on a daily disposable wear modality over a period of approximately one week.

DETAILED DESCRIPTION:
The study is a prospective, double masked (investigator and participant), bilateral, randomized, cross-over dispensing study, which evaluates somofilcon A (test lens) and etafilcon A (control lens).

ELIGIBILITY:
Inclusion Criteria:

* Subjects will only be eligible for the study if:

  1. Is at least 17 years of age and has full legal capacity to volunteer;
  2. Has read and signed an information consent letter;
  3. Is willing and able to follow instructions and maintain the appointment schedule;
  4. Habitually wears silicone hydrogel frequent replacement soft contact lenses, for minimum of 6-months;
  5. Is correctable to a visual acuity of 20/40 or better (in each eye) with the study lenses;
  6. Can be fit with study contact lenses with a power between - 0.50 and -10.00 DS;
  7. Demonstrates an acceptable fit with the study lenses;
  8. Habitually wears contact lenses for at least 8 hours per day, and willing to wear contact lenses for at least 12 hours a day in the study.

     Exclusion Criteria:
* Subjects will not be eligible to take part in the study if:

  1. Is participating in any concurrent clinical or research study;
  2. Has any known active* ocular disease and/or infection;
  3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
  4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
  5. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
  6. Is pregnant, lactating or planning a pregnancy at the time of enrolment (verbal confirmation at the screening visit);
  7. Is aphakic;
  8. Has undergone refractive error surgery;
  9. Is an employee of the Centre for Ocular Research & Education;
  10. Has participated in the BEAGLE (EX-MKTG-104) study.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-11-24 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Somofilcon A Then Etafilcon A: Subjects will be randomized to wear somofilcon A daily disposable lenses for one week and then switch to etafilcon A daily disposable lenses for one week.
  somofilcon A: Contact Lens etafilcon A: Contact Lens
- Etafilcon A Then Somofilcon A: Subjects will be randomized to wear etafilcon A daily disposable lenses for one week and then switch to somofilcon A daily disposable lenses for one week.
  etafilcon A: Contact Lens somofilcon A: Contact Lens
Period: First Intervention
Arm/Group | Somofilcon A Then Etafilcon A | Etafilcon A Then Somofilcon A
Started | 27 | 29
Completed | 27 | 29
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Somofilcon A Then Etafilcon A | Etafilcon A Then Somofilcon A
Started | 27 | 29
Completed | 26 | 29
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 56

OUTCOME MEASURES:

1. Primary Outcome: Lens Handling for Lens Insertion
Description: Lens handling for lens insertion (subjective rating; 0 - 10 integer scale, 0 - very difficult, 10 - very easy)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Somofilcon A: Subjects will be randomized to wear somofilcon A daily disposable lenses for one week.
  somofilcon A: Contact Lens
- Etafilcon A: Subjects will be randomized to wear etafilcon A daily disposable lenses for one week.
  etafilcon A: Contact Lens
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 9.3 (1.0) | 8.0 (1.9)

2. Primary Outcome: Lens Handling for Lens Insertion
Description: Lens handling for lens insertion (subjective rating; 0 - 10 integer scale, 0 - very difficult, 10 - very easy)
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 9.3 (1.2) | 7.9 (2.4)

3. Primary Outcome: Lens Handling for Lens Insertion
Description: Lens handling for lens insertion (subjective rating; 0 - 10 integer scale, 0 - very difficult, 10 - very easy)
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 9.2 (1.3) | 8.1 (2.3)

4. Primary Outcome: Lens Handling for Lens Insertion
Description: Lens handling for lens insertion (subjective rating; 0 - 10 integer scale, 0 - very difficult, 10 - very easy)
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 9.4 (0.8) | 8.1 (1.7)

5. Primary Outcome: Lens Handling for Lens Removal
Description: Lens handling for lens removal (subjective rating; 0 - 10 integer scale, 0 - very difficult, 10 - very easy)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 9.4 (1.0) | 9.3 (1.4)

6. Primary Outcome: Lens Handling for Lens Removal
Description: Lens handling for lens removal (subjective rating; 0 - 10 integer scale, 0 - very difficult, 10 - very easy)
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 9.2 (1.0) | 9.2 (1.3)

7. Primary Outcome: Lens Handling for Lens Removal
Description: Lens handling for lens removal (subjective rating; 0 - 10 integer scale, 0 - very difficult, 10 - very easy)
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 9.3 (1.0) | 9.1 (1.3)

8. Primary Outcome: Lens Handling for Lens Removal
Description: Lens handling for lens removal (subjective rating; 0 - 10 integer scale, 0 - very difficult, 10 - very easy)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 9.4 (0.7) | 9.3 (0.9)

9. Secondary Outcome: Lens Centration
Description: Lens Centration was measured on a scale of 0-3 (0 - optimal, 1 - slight decentration, 2- moderate decentration but not encroaching limbus, 3 - excessive & occasionally encroaching limbus)
Time Frame: Baseline (after 10 minutes of lens fitting)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 0.8 (0.5) | 0.7 (0.7)

10. Secondary Outcome: Lens Centration
Description: Lens Centration was measured on a scale of 0 - 3 (0-optimal, 1-slight decentration, 2-moderate decentration but not encroaching limbus, 3-excessive & occasionally encroaching limbus)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 0.7 (0.6) | 0.8 (0.6)

11. Secondary Outcome: Post-blink Movement
Description: Post-blink movement in primary gaze, in 0.1mm steps
Time Frame: Baseline (after 10 minutes of lens fitting)
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
millimeters | 0.3 (0.1) | 0.3 (0.1)

12. Secondary Outcome: Post-blink Movement
Description: Post-blink movement in primary gaze, in 0.1mm steps
Time Frame: 1 -week
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
millimeters | 0.3 (0.1) | 0.3 (0.1)

13. Secondary Outcome: Push-up Tightness
Description: Push-up tightness in primary gaze was measured using a scale 0-100 (5% steps) (0% = falls from cornea without lid support, 50% = optimum, 100% = no movement)
Time Frame: Baseline (after 10 minutes of lens fitting)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 51 (5) | 49 (5)

14. Secondary Outcome: Push-up Tightness
Description: as for outcome 13
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 52 (6) | 48 (7)

15. Other Pre Specified Outcome: Subjective Ratings of Comfort After Lens Insertion
Description: Subjective Ratings of Comfort After Lens Insertion was measured on a scale of 0-10 (0-Painful, 10- Can't feel the lenses).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 9.2 (1.0) | 8.7 (1.8)

16. Other Pre Specified Outcome: Subjective Ratings of Comfort After Lens Insertion
Description: as for outcome 15
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 9.1 (0.9) | 8.9 (1.4)

17. Other Pre Specified Outcome: Subjective Ratings of Comfort After Lens Insertion
Description: as for outcome 15
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 9.1 (1.2) | 8.6 (1.7)

18. Other Pre Specified Outcome: Subjective Ratings of Comfort After Lens Insertion
Description: as for outcome 15
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 9.2 (1.0) | 8.9 (1.3)

19. Other Pre Specified Outcome: Subjective Ratings of Comfort After Lens Insertion
Description: as for outcome 15
Time Frame: 1-Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Etafilcon A
Number analyzed (Participants) | 55 | 55
units on a scale | 9.0 (1.0) | 8.1 (1.8)

ADVERSE EVENTS:
Time Frame: From baseline till 1 -week for each type of lenses, up to 2 weeks total
Arm/Group | Somofilcon A | Etafilcon A
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 2/55 | 0/55
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somofilcon A (N=55) | Etafilcon A (N=55)
Conjuctival Staining (Eye disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT04195893/Prot_SAP_000.pdf